CLINICAL TRIAL: NCT00559299
Title: A Randomized, Single-blind, Placebo-controlled, 2 Part Study to Evaluate the Safety and Tolerability of GSK163090 at Single and Repeat Doses in Subjects With MDD
Brief Title: Patient Tolerability Study of GSK163090
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HTP110333
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Depressive Disorder, Major; Major Depressive Disorder (MDD)
Keywords: 163090; placebo-controlled; MDD; Depression; Tolerability; MDE
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — 1-(3-(2-(4-(2-methyl-5-quinolinyl)-1-piperazinyl)ethyl)phenyl)-2-imidazolidinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GSK163090

SUMMARY:
The purpose of this study is to determine the safety and tolerability of a new drug, GSK163090, which is being developed for the treatment of depression and anxiety disorders.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects between the ages of 18 - 65 years with a psychiatric diagnosis of a MDE associated with MDD according to DSM-IV-TR (296.2/296.3) whose symptoms are considered mild to moderate and have not been taking antidepressant medication at the time of screening and for at least 4 weeks prior to randomisation.
* If female, the subject is eligible to enter and participate in this study if she is not lactating and is of:

  1. Non-childbearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal [defined as one year without menses for women >45 years of age]); is surgically sterile [via hysterectomy and/or removal of the ovaries] or,
  2. Child-bearing potential, has a negative pregnancy test at both screen and baseline (prior to investigational product administration), and agrees to acceptable methods of contraception
* Body weight ≥ 50 kg and body mass index (BMI) between 18.5 - 35.0 kg/m2 inclusive.
* Capable of giving informed consent and can comply with the study requirements and timetable.
* Subjects have a HAM-D17 score > 18 and <25 at screening and baseline.
* The subject must be able to read, comprehend and record information.
* Non-smoker or light (< 10 cigarettes per day) smoker.
* Agree to abstain from alcohol for 24 hours prior to the start of dosing until collection of the final pharmacokinetic sample.

Exclusion Criteria:

* Subjects whose symptoms of the MDE are better accounted for by another diagnosis.
* As a result of any of the medical interview, physical examination or screening investigations the physician responsible considers the subject unfit for the study.
* The subject has a history of a drug reaction or other allergy which in the opinion of the physician responsible contraindicates their participation in the study.
* The subject is currently participating or has participated in a clinical trial with a new chemical entity or any investigational drug during the previous 2 months. In addition, the subject has not participated in clinical trials with more than 3 new chemical entities in the past 12 months.
* The subject has a screening ECG with parameters outside ranges defined in the protocol
* The subject has a pulse rate <45 or >100 bpm and/or a systolic blood pressure >150 and/or <90 and/or a diastolic blood pressure >90 and <50.
* History of long QT syndrome (personal or family) or other cardiac conduction disorder, or other clinically significant cardiac disease.
* The subject has any liver function test (LFT) elevated >1.5 times above the reference range at pre-study screening that remain elevated with a repeat LFT.
* Any other clinically significant laboratory abnormality.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John'sWort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and sponsor the medication will not interfere with the study procedures or compromise subject safety.
* Use of monoamine oxidase inhibitors (MAOI) and linezolid (antibiotic) for 1 month prior to first dose of study medication.
* Abuse of alcohol defined as an average weekly intake of greater than 21 units for males and 14 units for females or an average daily intake of greater than 3 units for males and 2 units for females. 1 unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* Consumption of grapefruit juice or grapefruit within 7 days prior to the first dose of study medication until collection of the last PK sample.
* The subject is unable to abstain from strenuous physical activity for 48 h prior to screening and follow up and for 48 h prior to and 48 h after each treatment period.
* Where participation in study would result in donation of blood in excess of 500 mL within a 90 day period
* An unwillingness of male subjects to abstain from, or use a condom during, sexual intercourse with pregnant or lactating women from the time of the first dose of study medication until 90 days following administration of the last dose of study medication
* OR
* An unwillingness of the male subject to use a condom/spermicide in addition to having their female partner use another form of contraception such as an IUD, oral contraceptives, injectable progesterone, subdermal implants or a tubal ligation if the woman could become pregnant from the time of the first dose of study medication until 90 days following administration of the last dose of study medication.
* Current or recent (within one year) gastrointestinal disease; a history of malabsorption, esophageal reflux, irritable bowel syndrome; frequent (more than once a week) occurrence of heartburn; or any surgical intervention (e.g., cholecystectomy) which would be expected to influence the absorption of drugs.
* Subjects who, in the investigator's judgement, pose a homicidal or serious suicidal risk, have made a suicide attempt within 6 months preceding screening or who have ever been homicidal.
* The subject has a history of a clinically significant abnormality of the neurological system (including dementia and other cognitive disorders or significant head injury) or any history of seizure (excluding febrile seizure).
* The subject has tested positive for hepatitis C antibody or hepatitis B surface antigen.
* The subject has tested positive for HIV.
* The subject has a past history of drug abuse or dependence according to DSM-IV TR criteria within the past 12 months or has tested positive for urine drugs of abuse at pre-study screening.
* The subject has any history of serotonin syndrome or in the investigator's judgement, a history of clinical significant intolerance to SSRIs.
* Subjects with a history of migraine headaches that respond to treatment with triptan medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GSK163090: Clinical laboratory, ECGs and vital signs assessments Questionnaire - DESS(Discontinuation Emergent Signs and symptoms) | All over 10 days post dose for Group 1 and over 3 weeks for subjects in groups 2 and 3.

SECONDARY OUTCOMES:
•Questionnaires •Prolactin, cortisol •PK parameters for GSK163090 | All over 10 days post dose for Group 1 and over 3 weeks for subjects in groups 2 and 3.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wichita, Kansas, United States